CLINICAL TRIAL: NCT01821014
Title: Satellite-supplementation of Medical Outreach Clinics: a Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bart M. Demaerschalk, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 13-000132
Record Dates: First submitted 2013-03-20; First posted 2013-03-29 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Telemedicine; Primary Health Care; Developing Countries; Diagnosis; Therapeutics
Keywords: Diagnostic concordance; Treatment concordance; patient satisfaction; physician satisfaction; Medical Outreach Clinics; Medical Brigades; Medical Missions; Telemedicine; Videoconference; diagnoses; treatments; Satellite Internet; VSAT; cross cultural telemedicine
MeSH Terms: conditions — Disease; Patient Satisfaction | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Telemedicine First (Experimental): Patients whose first physician visit during the clinic was using videoconference, a form of telemedicine, and whose second physician visit during the clinic was with a physician in-person.
  Interventions: Other: Telemedicine; Other: In-person physician interaction
- Telemedicine Second (Experimental): Patients whose first physician visit during the clinic was with a physician in-person, and whose second physician visit during the clinic was using videoconference, a form of telemedicine. This is the reverse order of visits of the "Telemedicine fist" arm.
  Interventions: Other: Telemedicine; Other: In-person physician interaction
- Two physician visits (Active Comparator): Patients who had two sequential visits with different in-person physicians.
  Interventions: Other: In-person physician interaction

INTERVENTIONS:
Other: Telemedicine — Patients undergo a detailed history and examination to the degree that is possible using the videoconference program, skype, a digital camera for high-resolution images, and an electronic stethoscope. A clinic volunteer aids with examination, translation and documentation.
  Other Names: Videoconference; Skype
  Arms: Telemedicine First; Telemedicine Second
Other: In-person physician interaction — Patients undergo a detailed history and examination by an in-person physician. A clinic volunteer aids with examination, translation and documentation, as needed.
  Other Names: in-person visit; in-person examination; in-person consultation

SUMMARY:
Much of the basic general medical care and chronic disease management in rural Honduras comes from groups of volunteers setting up temporary clinics run by volunteers. These clinics, also known as brigades, or medical missions, are often criticized for their lack of quality and the lack of follow-up, both of which stem, in part, from understaffing with volunteer physicians. This study is designed to assess if it is feasible, safe, and acceptable to treat patients in short-term mobile medical clinics in rural Honduras using US physicians connected with patients by videoconference.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent
* Non-emergent medical complaints
* At least 18 yrs in age

Exclusion Criteria:

* Pregnancy
* Mental Disability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2013-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Clinical Diagnoses | Same Day as clinic visit (less than 6 hours)
  The diagnoses resulting from the two physician visits will be compared and a cohen's kappa statistic will be calculated for diagnoses between the visits.
Recommended clinical treatments | Same Day as clinic visit (less than 6 hours)
  After each of a patient's two physician visits, the physician's resulting recommended treatments will be gathered for comparison between the two visits.

SECONDARY OUTCOMES:
Patient opinions of physician interactions | Immediately following physician interactions (less than 6 hours)
  Patients will receive a survey following each interaction with a doctor. These surveys cover communication, comfort and satisfaction.
Physician opinions of patient interactions | immediately following volunteer activities with the clinic (less than 48 hours)
  doctors will fill out a survey about their patient interactions after they complete their experience volunteering with the clinic.
Volunteer opinions of physician-patient interactions | immediately following experience with the clinic (Less than 48 hours)
  Volunteers who helped with physician interactions will receive a survey about their experience concerning physician patient communication, volunteer educational value and perceived value of the experience.

OTHER OUTCOMES:
Cost | One year (from pilot to completion of study)
  The costs of materials and services required to conduct the patient examinations will be collected to build an economic model and projected cost of scaling up the videoconference interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Bart Demaerschalk, MD/MSc, Principal Investigator — Mayo Clinic
Locations (1):
- Global Brigades, Tegucigalpa, Francisco Morazán Department, Honduras